CLINICAL TRIAL: NCT00141934
Title: Phase II Randomised, Double-Blind, Multicentre, Placebo-Controlled, Dose-Ranging, Parallel Group Study to Compare the Efficacy, Safety and Tolerability of 3 Strengths of AD 452 in Adults With Active RA Who Are Currently Taking Methotrexate.
Brief Title: A Multicentre Trial to Determine the Efficacy of AD 452 in RA Subjects.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sosei (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-AD452-022
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2007-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; RA; ACR20 endpoint; Tender/swollen joints; Improvement in pain; Health assessment questionnaire; Profile of mood states
MeSH Terms: conditions — Arthritis, Rheumatoid

INTERVENTIONS:
Drug: AD 452

SUMMARY:
AD 452 is a new drug which is being developed for use in adult patients with RA. It is believed that AD 452 may modify the underlying disease of RA as well as improving RA symptoms, and in order to establish its efficacy and safety, AD 452 is being tested in a 3 month study. Patients enrolled in this study will already be taking methotrexate for their RA and they will remain on methotrexate throughout the study. An earlier clinical study in 98 subjects with RA on stable background therapy investigated the pharmacokinetics, safety and tolerability of AD 452 taken for one month. The drug was well tolerated and no significant drug related adverse events were reported.

ELIGIBILITY:
Inclusion Criteria:

* Male/female age 18 -75
* RA diagnosed for at least 6 months
* Taking methotrexate for at least 6 months
* Must have at least 4 swollen/tender joints

Exclusion Criteria:

* Must not be pregnant/breastfeeding
* Must not have history of other inflammatory disorders
* Other conditions may lead to exclusion from the trial (e.g. Diabetes mellitus, malignant melanoma, HIV, active infection, hepatitis B/C, cardiac conduction disorders, hepatic/renal insufficiency, active depression/anxiety/psychosis/schizophrenia or convulsions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232
Dates: Start 2005-08

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Clinical Research of West Florida, Inc, Clearwater, Florida
  - Center for Rheumatology, Immunology and Arthritis, Fort Lauderdale, Florida
  - Ocala Rheumatology Research Center, Ocala, Florida
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - Advent Clinical Research Centers, Inc., St. Petersburg, Florida
  - Dept of Rheumatology, Columbia Medical Practice, Columbia, Maryland
  - Anderson and Collins Clinical Research, Inc., Edison, New Jersey
  - Station Avenue, Haddon Heights, New Jersey
  - Atlantic Coast Research LLC, Toms River, New Jersey
  - Rheumatic Disease Associates, Willow Grove, Pennsylvania